CLINICAL TRIAL: NCT01286649
Title: Randomized, Single-centre, Double-blind, Placebo-controlled, Phase I / IIa Study to Evaluate the Safety and Efficacy of Human Autologous Hair Follicle Dermal Sheath Cup Cells (DSCC) in Women and Men With Androgenetic Alopecia.
Brief Title: Safety and Efficacy Study of Human Autologous Hair Follicle Cells to Treat Androgenetic Alopecia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TrichoScience Innovations, Inc. (Industry)
Collaborators: Pharmalog Institut für klinische Forschung GmbH (PHARMALOG Institute for Clinical Research) (Unknown); PRA Health Sciences (Industry); Innovacell Biotechnologie AG (Industry); DatInf (Germany) (Unknown); The Hair and Skin Research and Treatment Center (Unknown)
Responsible Party: Sponsor
Organization: RepliCel Life Sciences, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: TS001-2009
Record Dates: First submitted 2011-01-18; First posted 2011-01-31 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Androgenetic Alopecia
Keywords: Alopecia; Alopecia, Androgenetic; Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Injection of verum and control (Other): Patients will receive randomized, blinded, injections of BOTH autologous hair follicle cells in medium (verum) and of medium alone (control) into two separate pre-defined treatment areas on their scalp.
  Interventions: Other: Human autologous hair follicle cells; Other: Cell medium

INTERVENTIONS:
Other: Human autologous hair follicle cells — Human autologous hair follicle cells suspended in cell medium
  Other Names: autologous hair follicle cells; hair follicle cells; verum
Other: Cell medium — Cell medium
  Other Names: control; placebo; cell transportation medium

SUMMARY:
The primary purpose of this study is to assess the safety of performing injections of human autologous hair follicle cells. The study will also measure the impact these injections will have on hair growth.

20 patients will be selected for participation in this study (10 males and 10 females) based on their health status, current/past medications, and ability to adhere to protocol-related requirements. All patients will have evidence of mild to moderate androgenetic alopecia (AGA) involving the vertex area of the scalp as defined by the Ludwig (female) or Norwood (male) scales.

At the first visit and after completing informed consent, patients provide a blood sample that will be tested for human immunodeficiency virus (HIV), hepatitis, and syphilis one week before having a biopsy from the back of their scalp. The provided scalp biopsy is then processed to isolate hair follicle cells which are then replicated. Patients return to the clinic for injections of their own replicated cells (autologous cells) in medium (verum) and medium alone (control) into two pre-selected treatment areas in their scalp. Assessments of the safety/tolerability of these injections will take place over the next 60 months both at in-clinic visits and telephone follow-up visits. At these visits patients will have their overall health assessed as subjective and objective assessments of the areas that were injected either with verum or control. During the first 24 months of follow-up, digital images will be taken of the scalp and of the two treatment areas injected with either verum or control. Furthermore at 6, 12, and 24 months post-injection, four patients (2 male and 2 female) at each time point will provide biopsies of the injection sites for histopathological analysis. At the 60 month time point, any patients not previously providing biopsies for histopathological analysis will provide biopsies. Total duration of patient participation is approximately 63 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the age of 18 and 55 years and in good health having evidence of mild to moderate androgenetic alopecia (AGA) involving the vertex area of the scalp. Female patients with androgenetic alopecia (AGA) characterized as vertex pattern type II or type III of the Ludwig Scale qualify for inclusion in this study. Males with androgenetic alopecia (AGA) involving the vertex area of the scalp, characterized as type III vertex- type VI on the Norwood Scale qualify for inclusion in the study.
2. Willingness to provide written informed consent for participation in the study, attend all study visits and complete all procedures required by this protocol.
3. The test areas (areas to be injected) are of uniform skin color without erythema, dark pigmentation or scars that may confound study results.
4. Willingness to forego the use cosmetic or medical products for hair loss throughout the course of the study.
5. Females must be post-menopausal for at least one year, surgically sterile, or, if of childbearing potential, using highly-effective methods of birth control. This method of contraception must be used at least 4 weeks prior to and during the entire duration of the clinical trial.

Exclusion Criteria:

1. Use of any product (medication or otherwise) which interferes with the hair growth cycle.
2. Any systemic medical treatment for hair loss (for example, Finasteride, Minoxidil, Dutasteride, or antiandrogens) within the last 12 months.
3. Start of contraception treatments containing chlormadinone or cyproterone acetate within the last 12 months.
4. Women who are pregnant or nursing.
5. Presence of any medical condition that influences the hair growth cycle (for example, alopecia areata, lichen planopilaris, lupus erythematosus, severe seborrheic eczema, psoriasis capitis or tinea capitis, untreated thyroid gland disease/goiter development, auto-immune diseases, etc.).
6. Any condition that, in the investigator's opinion would impact patient safety and/or a patient's ability to complete all study related procedures (for example, psychiatric illness, drug addiction, alcoholism, etc.).
7. Infection with human immunodeficiency virus (HIV), hepatitis, or syphilis.
8. Subjects diagnosed with cancer with or without chemotherapy treatment.
9. Sudden hair loss within the last 4 months unrelated to normal seasonal hair shedding or androgenetic alopecia (AGA).
10. Subjects in the process of or having completed surgical correction of hair loss in the past 24 months.
11. Participation in a cosmetic and/or pharmaceutical research study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2010-12; Primary Completion 2012-04 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
Incidence of local adverse events | six months post-injection
  Assessment of the local (at pre-selected treatment sites) safety profile of autologous hair follicle cells at six months compared to control as defined by adverse events (AEs) with respect to their causality, incidence, severity and seriousness

SECONDARY OUTCOMES:
Incidence of local adverse events | 12, 24 and 60 months post-injection
  Local (at pre-selected treatment sites) safety profile of autologous hair follicle cells at 60 months compared to control, defined by adverse events (AEs) with respect to their causality, incidence, severity and seriousness
Systemic adverse events | during 60-month observation period
Histopathological analysis | 6, 12. 24 and 60 months post-injection
  Biopsies are taken from treatment areas injected with verum and control from two male and two female patients (selected at random) at 6, 12, and 24 months post-injection. All patients not previously providing biopsies will do so 60 months post-injection. Biopsies sent to a blinded independent evaluator who will perform microscopic analysis of sections of the biopsies and provide reports detailing the difference between the biopsies of the two treatment areas per patient.
Complete safety profile | during 60-month observation period
  Analysis of the complete safety profile of study participants. Number and type of adverse events (AEs) will be listed per patient and as will reports from the patients selected to provide biopsies for histopathological analysis.
Hair Growth | 6 months post-injection and over 24-month observation period
  Hair growth will be assessed subjectively and objectively via a series of digital images taken from the scalp using standardized equipment. The following images will be taken: global scalp image pre shaving, global scalp image post-shaving (at select visits only), macroscopic images of each injection sites.

CONTACTS AND LOCATIONS:
Overall Officials: Nino Lortkipanidze, MD, PhD, Principal Investigator — Scientific Research Institute for Skin and Venereal Diseases
Locations (1):
- Scientific Research Institute for Skin and Venereal Diseases, Department of Dermatology, Tbilisi, Georgia

REFERENCES:
- See also: RepliCel Life Sciences, Inc. Website (Parent Co. of TrichoScience Innovations, Inc.) — http://www.replicel.com/